CLINICAL TRIAL: NCT05780229
Title: Effectiveness of Treatments of Massive Tears in the Shoulder Rotator Cuff, Assessed With Relevant Results for the Patient: A Mixed Methodology Study.
Brief Title: Effectiveness of Treatments for Massive Rotator Cuff Tears: Mixed Methodology.
Status: Active, not recruiting | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital Universitario Fundación Jiménez Díaz (Other); Parc Taulí Hospital Universitari (Other); Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: PI18/00152
Record Dates: First submitted 2023-02-21; First posted 2023-03-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Massive Rotator Cuff Tears; Shoulder Disease
Keywords: Mixed metholodgy; Massive Rotator Cuff Tears; Shoulder Disease; Comparative Effectiveness Research; Prosthesis; Arthroscopic Surgery; Conservative treatment
MeSH Terms: interventions — Conservative Treatment; Rehabilitation; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Massive Rotator Cuff Tears: Mixed Methodology: Phase 1: A theoretical sampling of maximum variation was carried out using a segmentation criterion, being the evaluation before or after the treatment in those patients who attended the visit in 5 Spanish hospitals.
  Phase 2: A consecutive sample of patients with massive rotator cuff tears, treated with conservative treatment, arthroscopy decompression surgery, or reverse prosthesis in 5 Spanish hospitals.
  Interventions: Procedure: Conservative treatment; Procedure: Arthroscopic Decompression Surgery; Procedure: Reverse Prosthesis; Drug: Pain-Relief Medication; Device: Reverse Prosthesis Device

INTERVENTIONS:
Procedure: Conservative treatment — The rehabilitation is based on restoring the balance of the shoulder joint. Aiming to diminish pain and restore function, pain control and inflammation are addressed during the firsts 3-6 weeks. Before week 3, pendulum movements are allowed to initiate mobilization of the shoulder joint. Aiming to gain (almost) complete shoulder joint mobility, a passive and active mobility exercise program is carried out. Lastly, the focus is on muscle reinforcement, performing a series of active exercises with weights or bands to exercise different muscles of the shoulder or the shoulder girdle.
  Other Names: Rehabilitation
Procedure: Arthroscopic Decompression Surgery — Arthroscopic decompression surgery of the rotator cuff tear consists of cleaning the subacromial space. The procedures that are sometimes performed to diminish pain may include, removing the inflamed bursa, releasing the long head of the biceps (if injured), or lightly burring the acromion bone under which the tendons slide.
Procedure: Reverse Prosthesis — The reverse prosthesis consists of shoulder articular joint replacement. The humeral head is sectioned, and, on the scapular side, a metal tray is placed, which is fixed with screws, and a metal half-sphere fixed to the metal tray. On the humeral side, a metal stem with a concave plastic component is placed to articulate with the metal half-sphere, allowing shoulder mobility without the need of rotator cuff muscles.
Drug: Pain-Relief Medication — In the reverse prosthesis procedure and arthroscopic decompression surgery, the pain-relief medication plan is a standard regimen for all patients, which can be modified as needed. This plan is based on 50mg of dexketoprofeno, 1g of paracetamol, and 100mg of tramadol.
Device: Reverse Prosthesis Device — In the reverse prosthesis procedure, a Delta III reverse shoulder prosthesis is applied. The original design was developed by Grammont in 1980's, and has 2 components: 1) a metal tray fixed with screws, and a metal half-sphere fixed to the metal tray, and 2) a concave polyethylene component.

SUMMARY:
The purpose of this study is: 1) to identify relevant treatment outcomes for people with massive rotator cuff tears of the shoulder joint, according to the experience of the affected people, to facilitate treatment shared decision-making during the specialist consultation in Spain; 2) to compare the effectiveness of conservative treatment, arthroscopic decompressive surgery and reverse prosthesis, in terms of patient's relevant outcomes and health-related quality of life.

DETAILED DESCRIPTION:
Primary Objectives:

Phase 1 (Qualitative):

1. To explore the perceptions, believes, experiences and coping strategies that are relevant results for people undergoing treatment of massive rotator cuff tears.
2. To identify the relevant outcomes for people with massive rotator cuff tears, and their experiences with the shared-decision making process.

Phase 2 (Quantitative):

a) To compare the effectiveness of conservative treatment, arthroscopic decompressive surgery and reverse prosthesis, in terms of patient's relevant outcomes and health-related quality of life.

Outline:

Phase 1:

A qualitative, interpretative, descriptive study with a hermeneutics phenomenological approach was conducted from an 'etic' (from phonetic) perspective. Through hermeneutical phenomenology it was intended to describe and understand the multiple meanings that people with massive rotator cuff tears give to their experience and the results they expect from their treatment. A theoretical sampling of maximum variation was carried out using a segmentation criterion, being the evaluation before or after the treatment in those patients who attended the visit of the specialist in Spain.

Phase 2:

This is a prospective observational study of a cohort with rotator massive cuff tears treated either with conservative treatment, arthroscopic decompressive surgery, or reverse prosthesis.

Participants were consecutively recruited in 5 Spanish hospital departments (located in two autonomous communities). Patients eligible for inclusion were: age 65-85 years, without previous surgical treatment in the affected shoulder, and complete rupture of the rotator cuff tendons, verified by magnetic resonance imaging. Patients were excluded if they have a neurological injury and/or an active infection.

Demographic and clinical characteristics at baseline are recorded at clinical sites and in the interview pretreatment, and include birthdate, sex, intervention, date of intervention, date of rehabilitation, chronic conditions, smoking status, employment status, and a question about the relevant outcome identified through the Phase 1.

Quality of Life questionnaires are administered centrally by telephone interviews before treatment and during follow-up at 6, 12 and 24 months after treatment. Quality of Life evaluations are gathered using computer-assisted telephone administration and include: (1) the Oxford Shoulder Score (OSS); and (2) the EuroQol-5 Dimension (EQ-5D-5L).

The sample size calculated to detect differences between groups (0.07 points in the EQ-5D-5L utility index, minimal important difference) was of 200 patients considering the three treatment groups, given a statistical power of at least 80% at a significance level of 5%, and lost to follow-up of 10%.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 85 years.
* No previous surgical treatment in the affected shoulder.
* Complete rupture of the rotator cuff tendons, verified by magnetic resonance imaging;

Exclusion Criteria:

* Neurological injury.
* Active infection.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with massive rotator cuff tears.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Relevant treatment outcome identified through the Phase 1 of the study. | Before treatment
  "Fend for yourself" was identified in the Qualitative Phase as a relevant outcome. It was captured through a question before treatment: "To what extent are you able to fend for yourself".
Change from baseline in relevant treatment outcome (identified through the Phase 1 of the study). | At 6, 12, and 24 months after treatment
  "Fend for yourself" was identified in the Qualitative Phase as a relevant outcome, and was captured through two questions: A) "To what extent were you able to fend for yourself before the injury?"; and B) "To what extent can you fend for yourself after treatment?".
Change in health-related quality of life measured with the Oxford Shoulder Score among shoulder treatments | Before and 6, 12, and 24 months after treatment
  The Oxford Shoulder Score (OSS) is a 12-item instrument assessing the impact of shoulder treatments and their outcomes. Response options for each OSS item are on a 4-level Likert scale, which ranges from 0 to 48, where higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Quality-Adjusted Life Years measured with the EuroQol-5 Dimensions | Before and 6, 12, and 24 months after treatment
  The EuroQol-5D Dimensions (EQ-5D-5L) is a generic econometric instrument that contains five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with five levels of severity in each dimension. From the possible combinations of scales and severity levels (3125 health states), a utility index is obtained, which ranges from 1 (perfect health) to negative values, 0 being the value attributed to death.
Ability to carry out normal daily activities measured with the Constant-Murley Score | Before and 6, 12, and 24 months after treatment
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters, which define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.

CONTACTS AND LOCATIONS:
Overall Officials: Montse Ferrer Forés, MD, Ph.D., Principal Investigator — IMIM-Hospital del Mar Medical Research Institute, 08003 Barcelona, Spain.; Carlos Torrens Cánovas, MD, Ph.D., Principal Investigator — Hospital del Mar, 08003 Barcelona, Spain,
Locations (6):
- Spain (6):
  - Parc Taulí Hospital Universitari, Sabadell, Barcelona
  - Health Services Research Group, IMIM-Hospital del Mar Medical Research Institute, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clínic, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Data processing complies with ethical principles and relevant national and international legislation (Reglamento General de Protección de Datos 2016/679 and Organic Law 3/2018, of December 5). The final data will only be accessible to people working on the study. No data used in the analyses and subsequent dissemination of the study results will contain any identifiable reference referring to the names of patients. Once the study is finished, the results will be communicated to the competent authorities, in accordance with local legislation.
  Data and associated documentation will be made available to users only under a data sharing agreement that provides for:
  * A commitment to use the data only for research purposes and not to identify any individual participant;
  * A commitment to protect data through the use of appropiate information technology;
  * A commitment to destroy or return the data after analyses are complete.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data and definitive documentation of the project will be stored centrally on virtual servers (up to 40 TB) and research storage infrastructures provided by the Hospital del Mar Medical Research Institute, during the lifetime of the project. Thereafter, the data will be kept for the recommended period of 20 years, as set out in the Medical Research Council's guideline "Personal Information in Medical Research" (section 7).
Access Criteria: Data sharing agreement among institutions.

REFERENCES:
- [Result] Barrufet C, Zamora V, Lizano-Barrantes C, Torrens C, Buron A, Calvo E, Peidro L, Miquel J, Barco R, Ferrer M. Relevant treatment outcomes for individuals aged 60 and older with massive rotator cuff tears: a qualitative study with 16 patients. Acta Orthop. 2025 Apr 14;96:322-330. doi: 10.2340/17453674.2025.43474. PMID 40223678